CLINICAL TRIAL: NCT02741804
Title: A Multi-domain Lifestyle Intervention Protocol to Detect Changes in Retinal Amyloid Among Individuals With Mild Cognitive Impairment
Brief Title: Lifestyle Intervention Program for Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ayesha Sherzai, MD, Staff Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 41387
Record Dates: First submitted 2016-04-07; First posted 2016-04-18 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Memory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BBH-1001 Brain Health Supplement (Active Comparator): Patients will be given supplement containing ingredients all approved by the FDA: Turmeric (125mg), fisetin (16.65mg), green tea leaf extract (17.5mg), EPA (75mg), DHA (150mg) and Vitamin D3 (250IU). Patients will take 4 softgels once per day for entire study duration (18 months).
  Interventions: Dietary Supplement: BBH-1001 Brain Health Supplement; Other: Lifestyle Intervention
- Brain Health Placebo (Placebo Comparator): Patients will be given a pill resembling the study supplement, but instead consisting of Soybean oil (608mg). Patients will take 4 softgels once per day for the entire study duration (18 months).
  Interventions: Other: Lifestyle Intervention; Dietary Supplement: Brain Health Placebo

INTERVENTIONS:
Dietary Supplement: BBH-1001 Brain Health Supplement — Treatment with supplement consisting of turmeric, fish oil, vitamin D and green tea extract OR placebo.
  Arms: BBH-1001 Brain Health Supplement
Other: Lifestyle Intervention — All patients will be given lessons on 6 areas of lifestyle: nutrition, physical activity, meditation, sleep hygiene, cognitive activity, and social activity.
Dietary Supplement: Brain Health Placebo — Treatment with placebo consisting of soybean oil
  Arms: Brain Health Placebo

SUMMARY:
The purpose of the Lifestyle Intervention Study is to investigate the influence of a micronutrient supplement in combination with a comprehensive lifestyle intervention program on retinal amyloid, among patients with Mild Cognitive Impairment (MCI). Patients will be placed on supplement or placebo throughout their 18-month study participation. Patients will also be given lifestyle training on nutrition, physical activity, cognitive and social activity, meditation and sleep, which have all been proven to positively affect cognition over time. Throughout their participation, patients' cognitive functioning will be monitored with comprehensive imaging, neuropsychological testing, blood testing and study compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years of age
* Experiencing memory, or cognitive problems

Exclusion Criteria:

* Patients < 55 years of age
* Previously diagnosed dementia; suspected dementia after clinical assessment by study physician at screening visit
* Mini Mental State Examination (MMSE) score less than 20 points
* Disorders affecting safe engagement in the intervention (e.g., malignant disease, major depression, psychiatric disease, symptomatic cardiovascular disease, revascularization within 1 year previously)
* Unable to safely change diet
* Patients without the means to visit the clinic on the assigned dates
* Patients that cannot comply with the data gathering needs of the study
* Severe loss of vision, hearing, or communicative ability
* Disorders preventing cooperation as judged by the study physician
* Coincident participation in another intervention trial
* Allergy to any ingredient in the supplement or placebo (i.e. soybean oil)
* Patients with gallstones due to possible interactions with turmeric
* Participants who are unable to provide clearance from their physician to participate in the physical activity training, as well as confirmed by Dr. Sherzai during the neurological exam.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in retinal amyloid burden, as measured by retinal amyloid scan. | baseline and 18 months
  Patients will be given a retinal scan at baseline, 6 months, 12 months and end of study (18 months). The retinal scanner is an device that measures the buildup of amyloid proteins in the brain via imaging of the eye. The change in amyloid buildup between each time point will be measured to determine effect of the interventions.

SECONDARY OUTCOMES:
Change in Neuropsychology | baseline and 18 months
  1) Cognitive performance measured by Neuropsychological Test Battery, evaluating several cognitive domains, which are sensitive measures for mild cognitive changes
Diagnosis of Dementia | baseline and 7-10 years
  2) Incidence dementia and Alzheimer's disease (according to standard criteria, NINCDS-ADRDA). An extended follow-up of at least 7-10 years is needed to investigate the effect of the intervention on this outcome.
Change in Neuroimaging | baseline and 18 months
  3) Neuroimaging via data review (structural and functional brain MRI and FDG-PET).
Change in Lab Results | baseline and 18 months
  4) Serum and plasma lab tests (inflammatory, metabolic, lipid and glucose metabolism, serum vitamin levels)
Change in Vascular Risk Factors | baseline and 18 months
  5) Vascular risk factor markers (blood pressure, blood glucose and HgA1c, lipid panel)

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Sherzai, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No